CLINICAL TRIAL: NCT04611906
Title: Evaluation of Small Vessel Disease by 3D-rotational Angiography
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. IP Yiu Ming Bonaventure, Specialist resident, Chinese University of Hong Kong
Other Study IDs: Crec 2020.386
Record Dates: First submitted 2020-10-27; First posted 2020-11-02 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Stroke, Acute; Stroke; Small Vessel Cerebrovascular Disease; Ischemic Stroke
Keywords: stroke; small vessel disease; 3D-rotational Angiography; Ischemic stroke
MeSH Terms: conditions — Stroke; Cerebral Small Vessel Diseases; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke patient: Patients who have acute cerebral ischemic symptoms attributed by cSVD can be recruited into this study. Eligible patients will be screened by Neurologists based on the inclusion and exclusion criteria. The time window for recruitment of the patient is 4 weeks from the qualifying stroke.

SUMMARY:
This study is aimed to elucidate the factors affecting the remodeling process of arteriolosclerosis under current practice recommendations. Such knowledge may improve the understanding of cerebral small vessel disease (cSVD) mechanism, define pharmacological therapy and suggest treatment target.

DETAILED DESCRIPTION:
Around 68 patients who have acute cerebral ischemic symptoms attributed by cSVD will be recruited. Stroke etiology will be determined by Neurologists based on clinical syndrome, vascular imaging features and concurrent cardiovascular risks. The time window for recruitment is 4 weeks from the qualifying stroke.

After an informed consent for the study, potential candidates will undergo a cranial MRI and MR angiography. Patients who are found to have acute or subacute lacunar infarcts (defined as an infarct diameter < 15mm) in the territories supplied by the lateral lenticulostriate arteries, i.e. internal capsule, putamen, external capsular or corona radiata, will proceed to a 3-Dimensional rotational angiography (3DRA) at baseline and in 12 months. All recruited patients will receive single antiplatelet agents and statin. Their cognition, mobility and treat cardiovascular risk factors based on 4 pre-specified goals (as elaborated in Study Procedures) will also be regularly reviewed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is Chinese ONLY
2. Patient is 30 to 85 years of age, inclusive.
3. Patients who have an acute lacunar infarct in diffusion-weighted MRI compatible with small vessel disease in territories supplied by the lateral lenticulostriate arteries without relevant intracranial atherosclerotic stenosis ≥60%.
4. Patient who has no contra-indication for the proposed imaging tests.
5. Patient who understands the purpose and requirements of the study, and has an informed consent.
6. Patient who has Modified Functional Ambulation Classification 4 or above.

Exclusion Criteria:

1. Stroke etiology uncertain or unrelated to small vessel disease, such as cardioembolism, Moyamoya disease, ICAD or primary angiitis of CNS.
2. Bleeding propensity: active peptic ulcer disease, major systemic hemorrhage within 30 days, thrombocytopenia (platelets <100 x 109/L), coagulopathy (INR >1.5).
3. A medical condition that would not allow the patient to adhere to the protocol or complete the study.
4. Patients with severe renal impairment.
5. Patients who are taking warfarin and non-vitamin K antagonist oral anticoagulants would also be excluded.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All ischemic stroke patients who have admitted to the Prince of Wales Hospital will be screened.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Morphological change | one year after recruitment
  The pre and post imaging in ischemic stroke patients by 3D-rotational angiography

CONTACTS AND LOCATIONS:
Overall Officials: Yiu Ming Bonaventure IP, MBChB, MRCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No